CLINICAL TRIAL: NCT04354805
Title: Administration of Chlorpromazine as a Treatment for COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Collaborators: Noha Mahmoud Nasreldin Hassan (Unknown)
Responsible Party: Principal Investigator, Ahmed Rezk, Clinical Instructor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medical
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Chlorpromazine

STUDY DESIGN:
Intervention Model Description: Single centred, single-blinded randomised controlled trial. All subjects from a population of interest will be randomly assigned to one of two groups, one group who is exposed to the intervention or a second group who receive the routine care in the hospital.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): The group of 50 patients are going to receive Chlorpromazine (oral dose of 50 mg/ day for 3 days then doubled to 100mg/day for further 11 days) every 24 hours for 14 days in addition to the convential treatment of COVID-19 according to the Egyptian Ministry of Health protocol.
  Interventions: Drug: Chlorpromazine
- Group B (No Intervention): A group of 50 patients control group who will recieve only the convential treatment of COVID-19 according to the Egyptian Ministry of Health protocol.

INTERVENTIONS:
Drug: Chlorpromazine — (Oral dose of 50 mg/ day for 3 days then doubled to 100mg/day for further 11 days)
  Other Names: Neurazine, Largactil
  Arms: Group A

SUMMARY:
In this study, defined cases of COVID-19 confirmed with PCR, with a mild, moderate or severe pneumonia will be treated with chlorpromazine. The improvement in clinical & laboratory manifestations will be evaluated in treated patient compared to control group.

DETAILED DESCRIPTION:
Introduction The COVID-19 pandemic has resulted in over 6 million confirmed infected cases worldwide and over 397,000 deaths as of June 8th, 2020 according to the World Health Organization. Currently, there is no specific medication for COVID-19, as there are different protocols of treatments that is not fully tested to prove its effectiveness by randomized control trials.

Due to high infectious potentials of COVID-19, all healthcare facilities are burdened out by an extra ordinary load which is reflected on the economy of the health sector. In Addition to public health measures like self-quarantine, isolation and social distancing, coming up with proved effective treatment for Covid-19 will help markedly in restoration of normal daily activity of people. In Egypt, public health measures are not much fruitful due to lack of people awareness to properly perform self-quarantine, economic burden for performing mass nasal swabs, some other factors such as uncertainty regarding the survival of the virus in air are subsequently adding much concern to the vast quarantine task.

Hence, the focus has now been directed toward evaluating and implementing other strategies like chemoprophylaxis and vaccination. In fact, the development of vaccine will take around two years as current human trials are being employed. Thus, the hope will be shifted towards the repurposing of an actually used drug to target the viral replication cycle.

Chlorpromazine is an antagonist of the dopamine receptor D2 (DRD2) and has been effectively and safely employed for over half a century in the treatment of psychiatric disorders (Adams, Awad, Rathbone, Thornley, & Soares-Weiser, 2014). The USA Food and Drug Administration approved the chlorpromazine as a first-generation antipsychotic. It is classified as a phenothiazine as its primary use is in the management of mental disorders to control mania and treatment of schizophrenia and it has several additional approved and off-label uses. Heart conduction abnormalities related to chlorpromazine use is only related to high doses. The most commonly reported signs and symptoms of acute toxicity are severe extrapyramidal reactions, hypotension, and sedation (Beckett, 2014).

Significance of the study Globally COVID-19 has led to large numbers of infection and death. In Egypt, number of confirmed cases increased above 30,000 according to the Egyptian Ministry of Health by 8th of June 2020. Furthermore, there is a change of the treatment protocol according to the severity of signs and symptoms aiming to decrease the load on the health facilities in Egypt.

The incubation period of COVID-19 is around 5.2 days at which the symptoms appears after (Li et al., 2020). The period from the onset of COVID-19 symptoms to death ranged from 1 week to 6 weeks with a median of 2 weeks (W., J., & F., 2020). This period is varied and can be determined according to the age and patient's immune system status. Patients > 70-years have a limited time compared to those under age of 70 (W. et al., 2020). The most symptoms at onset of COVID-19 illness are cough, fever and fatigue, shortness of breath in addition to sputum production, headache, dyspnea, diarrhea and lymphopenia (Huang et al., 2020; Ren et al., 2020; W. et al., 2020; Zhu et al., 2020). Clinically, a chest CT scan shows a diagnostic status of pneumonia, however, it is reflected clinically on patients showing acute respiratory distress syndrome, acute cardiac injury, and presence of grand-glass opacities that led to hypoxemia and death (Huang et al., 2020). At the molecular level, COVID-19 integration to the host cells requires active function of lysosome with a pH value from 4.5 to 5. This is the suitable pH for the bio-chemical reactions which leads finally to removal of the viral protein envelope and freedom of the viral genetic material for replication the molecular integration (Mindell, 2012).

Chlorpromazine has an alkaline effect on lysosomal pH. The significance in repurposing the chlorpromazine to target COVID-19 replication is due to the fact that an in-vitro dose of 0.82 μM leads to alkalization lysosome which is the lowest dose with no toxicity. The evidence of lysosomal pH alkalization was confirmed by a special fluorescent dye; LysoTracker Red1 DND-99 (LTR), which has been reported to accumulate in lysosomes by virtue of ionic trapping requiring acidic pH. The more LTR the more acidity of pH and vice versa, according to the study an evaluation was done after treatment of chlorpromazine with a concentration range from 200 μM to 0.82 μM. It was found that after 30 mins of chlorpromazine invitro treatment, there was a dose-dependent decrease of LTR staining (Lu, Sung, Lin, Abraham, & Jessen, 2017) . The lowest effective dose to transfer the invitro dose to in vivo calculated as follow:

(The desired dose x the molecular weight of the drug x average weight of patient in Kg)/1000

= (0.82 x 355 x 80 kg) / 1000 = 23.288 mg

Since the bioavailability of chlorpromazine is around 20-32% (Beckett, 2014; Boyd-Kimball et al., 2019). Thus, the dose might be required will be 100 mg. Since chlorpromazine is mostly metabolized by CYP2D6 in the liver, it would most likely exhibit patient dependent variable dose response. 100 mg dose could affect blood pressure thus cumulative dose will be considered. Initial start of dose will be 50 mg/ day for three days to be increased to100 mg/day till recovery. The toxicity of Chlorpromazine can occurs with a dose of 3000mg/day (Beckett, 2014). This is to further safeguard patients, clinical guideline and policy ought to be developed to provide ethical and legal framework for another use of chlorpromazine with COVID-19, also to follow the guidelines and institutional policies for using this medication within the hospitals.

Moreover, clinicians and Care givers can add chlorpromazine to the protocol of medical treatment for COVID-19 by providing evidence-based and comprehensive recommendation on the potential benefits, risks and related safety issues. The investigator believed that study will give the clinician an evidenced based practice to control COVID-19 replication using chlorpromazine. Although the literature revealed a possible hypotension effect from high doses of chlorpromazine, there are still risks of slight hypotension occurrence from low dose due to the nature of drug.

Lack of drugs for treatment of COVID-19 is adding much value to the significance and the originality of this study. The investigator aims at providing an evidence base for the effect of chlorpromazine on clinical picture progress of COVID-19 patients.

Aim of the study:

The study aims to evaluate the effect of chlorpromazine on reduction of illness severity among COVID-19 patients.The improving clinical outcomes and reducing the need for ventilator support will be evaluated in treated patient compared to control group. Approximately 100 participants hospitalized with COVID-19 in Cairo University hospitals will be enrolled into this study.

Research hypothesis:

In order to fulfill the aim of the study, the following research hypothesis will be postulated:

H. The chlorpromazine administration leads to reduction of illness severity estimated by WHO ordinal scale over time. Primary objective will be assessed by scale score at day 0, 3, 7, 11 and 15 from date of randomization.

Sub hypotheses:

H1. The chlorpromazine administration affects temperature mean scores compared to control group who receive the routine regimen among COVID-19 patients H2. The chlorpromazine administration affects heart rate mean scores compared to control group who receive the routine regimen among COVID-19 patients.

H3. The chlorpromazine administration affects respiratory rate mean scores compared to control group who receive the routine regimen among COVID-19 patients.

H4. The chlorpromazine administration affects oxygen saturation mean scores compared to control group who receive the routine regimen among COVID-19 patients H4. The chlorpromazine administration affects need for oxygen compared to control group who receive the routine regimen among COVID-19 patients.

H5.The chlorpromazine administration affects hospital stay time mean scores compared to control group who receive the routine regimen among COVID-19 patients.

H6. The chlorpromazine administration affects chest CT patches scores compared to control group who receive the routine regimen among COVID-19 patients.

H7. The chlorpromazine administration affects D Dimer mean scores compared to control group who receive the routine regimen among COVID-19 patients.

H8. The chlorpromazine administration affects Lymphocyte count mean scores compared to control group who receive the routine regimen among COVID-19 patients.

H9. The chlorpromazine administration affects C-reactive protein (CRP) mean scores compared to control group who receive the routine regimen among COVID-19 patients.

H10. The chlorpromazine administration affects Lactate dehydrogenase (LDH) mean scores compared to control group who receive the routine regimen among COVID-19 patients.

H11. The chlorpromazine administration affects S ferritin mean scores compared to control group who receive the routine regimen among COVID-19 patients.

H12. The chlorpromazine administration affects arterial blood gases mean scores compared to control group who receive the routine regimen among COVID-19 patients.

H13. The chlorpromazine administration affects temperature mean scores compared to control group who receive the routine regimen among COVID-19 patients H14. The chlorpromazine administration affects Creatine Phosphokinase (CPK) mean scores compared to control group who receive the routine regimen among COVID-19 patients.

H15. The chlorpromazine administration affects time for negative PCR of COVID-19 compared to control group who receive the routine regimen among COVID-19 patients.

Methods

Research design:

Single centred, single-blinded randomised controlled trial. All subjects from a population of interest will be randomly assigned to one of two groups, one group who is exposed to the intervention or a second group who receive the routine care in the hospital.

Settings This study will be conducted at New EL Kasr Al Aini hospital isolation wards. New EL Kasr Al Aini is Cairo University affiliated hospital. The COVID-19 patients are referred for isolation unit who receive COVID-19 protocol of treatment according to the Egyptian Ministry of Health.

Sample:

A convenient sample of patients with COVID-19 patients will be randomly assigned to two groups; study and control group. Data will be collected over a duration of 14 days, considering that patients will not be less than 100 patients.

Description of the experimental work (Chlorpromazine administration) The study group will be chosen to match the inclusion criteria, after that the investigator will obtain a written consent from patients who are willing to participate in the study. Randomization of subjects followed by a baseline laboratory , clinical data and illness severity score according to WHO ordinal scale will be recorded for both groups, then an initial dose of 50 mg of chlorpromazine hydrochloride orally once daily at night for three days to be doubled to 100mg / day till recovery criteria are met with maximum of 14 days. Evaluation of laboratory and clinical findings will start at day 0, 3, 7, 11 and 15 from day of randomization.

Ethical consideration Once the protocol is granted from Ethics and Research committee, an official permission will be taken from hospital administrators. Also; each patient will be informed about the purpose of the study and its importance. The investigator will confirm with the patients that sharing in this study is on voluntary bases. They have the right to withdraw from research without any penalty and this will not affect the provided routine care. Anonymity and confidentiality are assured through coding the data. The study subjects will be informed that the data will not be reused in another research without their permission. Informed consent will be taken from the patients who accept to be included in the study.

Procedure:

Upon receiving the formal approval to conduct the study, an official permission will be obtained from hospital director to proceed with the proposed study. The study participants will be selected according to the inclusion criteria, then the investigator will obtain a written consent from participants who are willing to participate in the study. Participants will be randomly assigned into study and control group. Both groups will receive the routine regime of medical treatment, During the implementation, baseline clinical, laboratory data and illness severity score will be recorded for both groups. However, the study group will receive initially a dosage of 50 mg of chlorpromazine hydrochloride orally once daily at night for duration of three days. Dose will be doubled to 100 mg/ day till recovery criteria are met with maximum of 14 days. The dose is calculated according to the bioavailability and the lowest effective required dose to rich the cells which should be not less than 0.82 uM (Lu et al., 2017). Finally, both groups will be monitored utilizing the tool sheets, any complications will be noted and will be reported for both groups. The investigator will record the values of assessment of patient at which heart rate and peripheral oxygen saturation will be assessed by pulse oximetry, respiration will be counted by the investigator and blood pressure will be assessed by digital or mercury sphygmomanometer. Recording of laboratory and clinical data will be done.

Data analysis:

Obtained data will be tabulated, computed and analyzed using Statistical Package for Social Science (SPSS) program version 21. Descriptive as frequency, mean, standard deviation…etc., in addition to inferential statistics as T.test and ANOVA will be utilized to analyze data pertinent to the study. Level of significance will be at P ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Adult conscious male and female (non-pregnant, non-breast feeder), level of consciousness is assessed by Glasgow Coma Scale ≥ 13.
2. Diagnosed initially with COVID-19 confirmed with PCR prior to any interference.
3. Follow the treatment regimen for COVID-19 according to The Ministry of Health in Egypt.

   Exclusion criteria:
4. Patients having allergy to chlorpromazine which will be assessed by asking the patient or relative.
5. Patients with hypotension(<90/60mmHg).
6. Pregnant and breast feeder female patients.
7. Hepatic patients.
8. Patients already receiving chlorpromazine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 2 weeks
  In the current study, the clinical improvement will be determined by:
  1. Temperature
  2. Heart rate (pulse)
  3. Respiratory rate
  4. Oxygen saturation
  5. Need for oxygen
  6. Hospital stay time.
  7. CT lung involvement at day 0 and day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Rezk, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: September 2020 to December 2020
Access Criteria: Direct contact with the investigator